CLINICAL TRIAL: NCT00769678
Title: Biventricular Pacing and Stimulation of the Diaphragm in Patients With Severe Heart Failure Following Heart Surgery (Epiphrenic II Pilot Trial)
Brief Title: Stimulation of the Diaphragm in Patients With Severe Heart Failure Following Heart Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Luzerner Kantonsspital (Other)
Collaborators: Inovise Medical (Industry)
Responsible Party: Principal Investigator, Prof. Paul Erne, Prof. Paul Erne, Luzerner Kantonsspital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Epiphrenic II Pilot Trial
Record Dates: First submitted 2008-10-03; First posted 2008-10-09 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-04

CONDITIONS: Heart Failure
Keywords: Biventricular Pacing
MeSH Terms: conditions — Heart Failure

ARMS (1):
- Stimulation of diaphragm (Active Comparator)
  Interventions: Device: Stimulation of the diaphragm

INTERVENTIONS:
Device: Stimulation of the diaphragm — Stimulation of the diaphragm using an electrode

SUMMARY:
This study examines whether a permanent stimulation of the diaphragm improves left ventricular function in patients with severe heart failure following heart surgery.

DETAILED DESCRIPTION:
Previous studies have shown that temporary stimulation of the diaphragm using an electrode to the phrenic nerve reduces electrical mechanical activation time (EMAT) and improves left ventricular function. This study examines whether patients with severe heart failure, who require permanent biventricular pacing after heart surgery, may benefit from an additional permanent electrode that stimulates the diaphragm. Heart function is assessed by echocardiography and acoustic cardiography (Audicor, Inovise Medical Inc., Portland, USA).

ELIGIBILITY:
Inclusion Criteria:

* Patients following open heart surgery who need permanent pacing

Exclusion Criteria:

* Patients with fast changing need of vasopressors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2008-10; Primary Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Left ventricular ejection fraction | One day

SECONDARY OUTCOMES:
Brain natriuretic peptide (BNP) | One day
6-minutes walking distance | One day
NYHA functional class | One day

CONTACTS AND LOCATIONS:
Locations (1):
- Kantonsspital Luzern, Lucerne, Canton of Lucerne, Switzerland

REFERENCES:
- [Derived] Beeler R, Schoenenberger AW, Bauer P, Kobza R, Bergner M, Mueller X, Schlaepfer R, Zuber M, Erne S, Erne P. Improvement of cardiac function with device-based diaphragmatic stimulation in chronic heart failure patients: the randomized, open-label, crossover Epiphrenic II Pilot Trial. Eur J Heart Fail. 2014 Mar;16(3):342-9. doi: 10.1002/ejhf.20. Epub 2013 Dec 6. PMID 24464736